CLINICAL TRIAL: NCT06536114
Title: Efficacy of a Criteria Based Clinical Pathway for Rehabilitation of Shoulder Injuries
Acronym: CRISP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Collaborators: Brooke Army Medical Center (U.S. Federal Agency); Congressionally Directed Medical Research Programs (U.S. Federal Agency); Henry M. Jackson Foundation for the Advancement of Military Medicine (Other); The Geneva Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMCSD.0024.0048
Record Dates: First submitted 2024-07-31; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Shoulder Pain; Shoulder Injuries
Keywords: shoulder; return-to-duty; physical therapy; rehabilitation
MeSH Terms: conditions — Shoulder Pain; Shoulder Injuries | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: multi-site, single-blinded, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will not be a physical therapist and thus not involved with the participant's medical treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Criteria-based Rehabilitation for Injured Shoulders Paradigm (CRISP). (Experimental): The CRISP group will undergo physical therapy treatment, directed by a research physical therapist, including both supervised physical therapy and a guided home exercise program.
  Interventions: Other: CRISP: Criteria-Based Approach for the Rehabilitation for Non-Operative Shoulder Injuries
- Standard of Care (Active Comparator): The standard of care group will serve as the control arm and complete a period of physical rehabilitation under the supervision of a Military Health System physical therapist without study-specific guidance or interventions.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: CRISP: Criteria-Based Approach for the Rehabilitation for Non-Operative Shoulder Injuries — The CRISP group will undergo physical therapy treatment, directed by a research physical therapist, including both supervised physical therapy and a guided home exercise program. This approach has three phases: stabilization, to facilitate joint protection; strength and endurance, to optimize functional capacity; and power, to prepare the Service member for returning to previous level of duty.
  Arms: Criteria-based Rehabilitation for Injured Shoulders Paradigm (CRISP).
Other: Standard of Care — The Standard of Care group will serve as the control arm and complete a period of physical rehabilitation under the supervision of a Military Health System physical therapist without study-specific guidance or interventions.
  Arms: Standard of Care

SUMMARY:
The goal of this clinical trial is to compare the current standard of care for rehabilitation of non-operative shoulder injuries to a novel, criteria-based approach (CRISP). Additionally, this study will identify factors which contribute to return to duty readiness. The main questions it aims to answer are:

* Are there differences in patient reported outcomes between participants who undergo the criteria-based rehabilitation program versus the standard of care for shoulder injuries?
* Are there differences in clinical measures (strength, etc.) between participants who undergo the criteria-based rehabilitation program versus the standard of care for shoulder injuries?
* Are there clinical or rehabilitation factors, or participant characteristics, that contribute to return to duty readiness?

Participants will be randomized to either complete their rehabilitation per the standard of care with a physical therapist in a Military Treatment Facility or complete the CRISP program with a research physical therapist. Participants will:

* Attend physical therapy for a non-operative shoulder injury
* Attend initial and final clinical assessments at the clinic
* Complete patient reported outcomes at 1-, 3-, 6- and 12-month timepoints

DETAILED DESCRIPTION:
Without a data-driven pathway to assess and rehabilitate shoulder injuries, clinicians may be using time rather than criteria to guide rehabilitation and clearance for return to duty. Delayed return to duty and subsequent injury or surgery contribute to time lost from duty, negative financial implications for the Military Health System, and adversely affect Service members' mental health and quality of life. Therefore, we propose a study determining the optimal treatment progression to reduce unnecessary variability in management of non-operative of shoulder injuries for Service members through a phased, criteria-based clinical pathway: Criteria-based Rehabilitation for Injured Shoulders Paradigm (CRISP). Additionally, this study will identify factors which contribute to return to duty readiness.

To demonstrate the benefits of the CRISP program, we will determine the differences in physical, psychological, and quality of life patient-reported questionnaires, and clinical assessments of shoulder strength and function between the novel criteria-based rehabilitation program and the current standard of care for Service members with non-operative shoulder injuries within the Military Health System. To accomplish this, we will conduct a multi-site, single-blinded, randomized controlled trial in active duty Service members seeking care for a non-operative shoulder injury referred to physical therapy. We will recruit 250 Service members from the Naval Medical Forces (Pacific Region) and Brooke Army Medical Center/Center for the Intrepid. Participating Service members will complete clinical assessments and questionnaires at initial and final assessments; additionally, a link will be sent to participants to fill out questionnaires virtually at 1-, 3-, 6-, and 12-month time intervals. The CRISP group will undergo physical therapy treatment, directed by a research physical therapist, including both supervised physical therapy and a guided home exercise program. This approach has three phases: stabilization, for joint protection; strength and endurance, for functional capacity; and power, to prepare the Service member for returning to previous level of duty. The standard of care group will serve as the control arm and complete a period of physical rehabilitation under the supervision of a Military Health System physical therapist without study-specific guidance or interventions. To our knowledge, this is the first study to compare a criteria-based exercise intervention approach to the usual standard of care for the conservative treatment of shoulder injuries as well as identifying factors which contribute to RTD readiness.

Without using a data-driven pathway to assess and rehabilitate shoulder injuries, Service members may experience a potential delay in returning to their previous military occupational specialty or deployability, and residual impairments may persist. In turn, this could lead to a higher incidence of re-injury or referral to surgical intervention. In the near-term, the findings from this study will enhance individual patient care within the MHS, accelerating return to duty for our Service members and with fewer physical limitations. We also anticipate our findings will help identify the predictors of shoulder function and return to duty readiness. This study's findings will directly influence patient care by elucidating which treatment paradigm optimizes shoulder function in Service members, ultimately leading to improvements in quality of life for Service members, reducing time lost from injuries, as well as maximizing Service members' readiness, unit cohesion, and mission accomplishment.

ELIGIBILITY:
Inclusion Criteria:

* Active-duty Service members over the age of 18 who are seeking medical attention for shoulder pain or injury will be recruited to participate in this study.

Exclusion Criteria:

* The exclusion criteria include individuals who have sustained cervical or thoracic spine injury in the past year; an upper extremity or spine injury within the past year and have not been cleared to perform their previous duty requirements; a diagnosis of adhesive capsulitis; individuals referred to post-operative rehabilitation for the shoulder; individuals who are scheduled for shoulder surgery within the following 12 weeks; pain originating from a body region other than shoulder or is non-orthopaedic in nature; individuals who have sustained an upper extremity limb loss; individuals pending a medical evaluation board, discharge from the military, or pending litigation for an injury.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Penn Shoulder Score | Initial and final clinical study assessments; 1-, 3-, 6- and 12-months post-randomization
  Patient-reported outcome with shoulder pain, satisfaction, and function subscales

SECONDARY OUTCOMES:
Referral to Surgical Intervention | 3-, 6-, 12- months
  Participant was referred to surgical invention for their shoulder injury.
Patient-Reported Outcomes Measurement Information System (PROMIS®) | Initial and final clinical study assessments; 1-, 3-, 6- and 12-months post-randomization
  Patient-reported outcome measuring physical, mental, and social health among individuals with various chronic conditions.
Optimal Screening for Prediction of Referral and Outcome- Yellow Flag (OSPRO-YF) | Initial and final clinical study assessments; 1-, 3-, 6- and 12-months post-randomization
  The OSPRO-YF is a 10-item screening tool which incorporates several psychosocial domains, namely, mood, fear avoidance, and positive affect-coping.
Military Orthopaedics Tracking Injuries and Outcomes Network (MOTION) Readiness Rehab Questionnaire | Initial and final clinical study assessments; 1-, 3-, 6- and 12-months post-randomization
  The Readiness Rehab Questionnaire assesses deployment readiness, containing questions including, "if called for a 6 month deployment today, my confidence to travel to/within a combat zone, carry/wear/use all required equipment and/or weapon, and perform required military duties for the duration of the 6 month deployment is:" and "my confidence to do my specific military duties with well managed pain is:__", both scored on 0-100 scales.

CONTACTS AND LOCATIONS:
Overall Officials: Marisunta Pontillo, PhD, Principal Investigator — Extremity Trauma and Amputation Center of Excellence, Defense Health Agency
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barber P, Pontillo M, Bellm E, Davies G. Objective and subjective measures to guide upper extremity return to sport testing: A modified Delphi survey. Phys Ther Sport. 2023 Jul;62:17-24. doi: 10.1016/j.ptsp.2023.05.009. Epub 2023 May 27. PMID 37300969
- [Background] Owens BD, Dawson L, Burks R, Cameron KL. Incidence of shoulder dislocation in the United States military: demographic considerations from a high-risk population. J Bone Joint Surg Am. 2009 Apr;91(4):791-6. doi: 10.2106/JBJS.H.00514. PMID 19339562
- [Background] Pontillo M, Sennett BJ, Bellm E. USE OF AN UPPER EXTREMITY FUNCTIONAL TESTING ALGORITHM TO DETERMINE RETURN TO PLAY READINESS IN COLLEGIATE FOOTBALL PLAYERS: A CASE SERIES. Int J Sports Phys Ther. 2020 Dec;15(6):1141-1150. doi: 10.26603/ijspt20201141. PMID 33344031
- [Background] Pontillo M, Spinelli BA, Sennett BJ. Prediction of in-season shoulder injury from preseason testing in division I collegiate football players. Sports Health. 2014 Nov;6(6):497-503. doi: 10.1177/1941738114523239. PMID 25364482